CLINICAL TRIAL: NCT04057430
Title: Effectiveness of the GumChucks® Flossing System Compared to String Floss for Interdental Plaque Removal in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nini Chaichanasakul Tran, DDS, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GumChucksEfficacy
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Gingivitis; Plaque
Keywords: Interdental plaque; Flossing aid; Children; Gingival inflammation
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- String floss (Active Comparator)
  Interventions: Device: String floss
- Gumchucks floss (Experimental)
  Interventions: Device: GumChucks

INTERVENTIONS:
Device: GumChucks — GumChucks® is an innovative flossing system resembling mini nunchucks. The two-handle design eliminates the need to wrap the floss around fingers, and a proper flossing technique is facilitated by the nature of its curved shaped.
  Arms: Gumchucks floss
Device: String floss — Traditional string floss used in this study was Oral-B Glide® Pro-Health Original Floss
  Arms: String floss

SUMMARY:
This study evaluates the interdental plaque removal efficacy, flossing speed, and reduction in gingival inflammation of a new flossing system (GumChucks®) compared to string floss, and to assess preference between the two flossing products in children, parents, and dentists.

ELIGIBILITY:
Inclusion Criteria:

* healthy children aged 4-15 years, who were not on any type of medication
* presence of at least 4 posterior interdental contacts
* ability to follow verbal and/or written instruction
* availability for a 4-week study period
* one parent or legal guardian of each included child participant.

Exclusion Criteria:

* had antibiotics within the last 6 months
* are pregnant.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-12-10 (Actual); Primary Completion 2017-02-26 (Actual); Study Completion 2017-02-26 (Actual)

PRIMARY OUTCOMES:
Interdental plaque score - after first use | Baseline and Day 1
  Interdental plaque scores were recorded after the teeth were stained with plaque disclosing solutions (GUM® Red-Cote®) for 30 seconds followed by a water rinse. Interdental plaque was scored either presence or absence at 4 sites of each tooth (mesio-buccal, disto-buccal, mesio-lingual, and disto-lingual).
  Score of 0 = If disclosing solution shows no visible plaque at the site Score of 1 = if disclosing solution shows the presence of any plaque between interproximal contact and the respective line angle of that site.
  The total interdental plaque score for each participant is the sum of all sites stained positive with disclosing solution.
Interdental plaque score - after 4 weeks of usage | Baseline and 4 weeks
  Interdental plaque scores were recorded after the teeth were stained with plaque disclosing solutions (GUM® Red-Cote®) for 30 seconds followed by a water rinse. Interdental plaque was scored either presence or absence at 4 sites of each tooth (mesio-buccal, disto-buccal, mesio-lingual, and disto-lingual).
  Score of 0 = If disclosing solution shows no visible plaque at the site Score of 1 = if disclosing solution shows the presence of any plaque between interproximal contact and the respective line angle of that site.
Gingival index - after 4 weeks of usage | Baseline and 4 weeks
  Gingival inflammation was assessed using the gingival index where the scores were taken of the buccal and lingual margins of the interdental papillae adjacent to interdental contacts with the following scoring system:
  0 = absence of inflammation
  1. = mild inflammation: slight change in color, little change in texture
  2. = moderate inflammation: moderate erythema/edema, bleeding on pressure
  3. = severe inflammation: severe erythema/edema, tendency to spontaneous bleeding, ulceration The gingival index score of each participant is the sum of all scores divided by the total numbers of buccal and lingual interdental papillae sites
Flossing speed | Day 1
  The total time for a participant to floss all interdental contacts was measured in seconds.

SECONDARY OUTCOMES:
Floss preferences by children, parents and dentists | Day 1
  Preferences of child participants, their parents and dentists toward the use of GumChucks® in comparison to string floss was measured by a 5-point Likert scale questionnaire. Child participants and their parents completed questionnaires after using both flossing products, while dentists completed questionnaires after viewing the video and/or live demonstration of GumChucks® usage on a model of the oral cavity.